CLINICAL TRIAL: NCT02293135
Title: Evaluation of the Action of the Stendo Pulsating Suit on Peripheral Microcirculation and on Endothelial Function in Diabetic Patients Without Complication
Brief Title: Evaluation of Stendo Pulsating Suit on Microcirculation and Endothelial Function in Diabetic Patients
Acronym: Diabete_1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stendo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00961-46
Record Dates: First submitted 2014-11-07; First posted 2014-11-18 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes ; endothelium stimulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Verum Stendo session on V1 and Phantom Stendo session on V2
  Interventions: Device: Verum Stendo session on V1 and Phantom Stendo session on V2
- Group 2 (Experimental): Phantom Stendo session on V1 and Verum Stendo session on V2
  Interventions: Device: Phantom Stendo session on V1 and Verum Stendo session on V2

INTERVENTIONS:
Device: Verum Stendo session on V1 and Phantom Stendo session on V2 — On the firt V1 visit, the patient will receive the verum Stendo session ; then on V2 visit ((V1 + 13 days +/- 2), the patient will receive the verum Stendo session On the firt visit, V1 the patient will have a phantom Stendo session (no pressure will be applied)
  Arms: Group 1
Device: Phantom Stendo session on V1 and Verum Stendo session on V2 — On the firt V1 visit, the patient will have a phantom Stendo session (no pressure will be applied) ; then on V2 visit ((V1 + 13 dayx +/- 2), the patient will receive the verum Stendo session
  Arms: Group 2

SUMMARY:
The action of one Stendo pulsating suit session will be evaluated on 16 type 2 diabetic patients referred on the diabetic consultations. The effects of one Stendo pulsating suit session system will be assessed on the peripheral cutaneous microcirculation and on endothelial functions

DETAILED DESCRIPTION:
The role of the endothelium in micro-vascular system is mediated by synthesis and release of numerous substances that act on the smooth muscle fibers. The release of these products is modulated, in turn, by various circulating molecules, by autonomic nervous system and by local mechanical factors such as shear stress.

The type 2 diabetes leads to early vascular redesign with the onset of endothelial dysfunction and the worsening of the arterial stiffness.

These anomalies, well correlated with the cardiovascular risks, are currently investigated in the department of Endocrinology, Diabetes, and Nutrition at the Jean Verdier Hospital. The analysis methods allow identifying early modifications in response to various drugs, nutritional or physical stimuli.

The aim of this study is therefore to evidence a peripheral microcirculation and endothelial function improvement in type 2 diabetic patient in comparison to a cross-over control session.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patient
* Diagnosis of diabetes > 1 year
* HBA1c between 6 and 8,5
* Treated with oral anti-diabetic, insulin and/or incretins which can be stayed unchanged during the 2-week study

Exclusion Criteria:

* Type 1 diabetic Patient
* Antecedent of cardiomyopathy, cardiac ischemia or valvulopathy
* Severe kidney failure
* Non controlled hypertension (> 160/100mm Hg)
* Cardiac arrhythmia
* Severe respiratory failure
* Patient with an advanced obstructive arterial disease
* Patient with a recent and progressive deep venous thrombosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Peripheral microcirculation measured using Laser Doppler flowmetry | 30 minutes after the end of the Stendo session
  Change in % of the peripheral cutaneous microcirculation using laser Doppler flowmetry after one Stendo pulsating suit session

SECONDARY OUTCOMES:
Arterial stiffness | 10 minutes after the end of Stendo session
  Change of arterial stiffness using an applanation tonometry device after one Stendo pulsating suit session; Augmentation Index and sub-endocardial viability ratio will also be assessed
Heart Rate Variability (HRV) | 15 minutes after the end of Stendo session
  HRV is calculated from continuous noninvasive arterial pressure records and continuous high resolution 3-lead, 6channel ECG records
Endothelium-dependant microvascular flow after local acetylcholine iontophoresis | 35 minutes after the end of Stendo session
  3 minutes Area Under Curve (AUC) of the peripheral microcirculation using Laser Doppler flowmetry
Reactive Hyperemia Index (RHI) | 45 minutes after the end of Stendo session
  RHI is the post-to-pre occlusion Peripheral Arterial Tone (PAT) signal ratio in the occluded arm, relative to the same ratio in the control arm

CONTACTS AND LOCATIONS:
Overall Officials: Paul VALENSI, Professor, Principal Investigator — Hôpital Jean Verdier
Locations (1):
- Hôpital Jean Verdier, Service d'Endocrinologie Diabétologie Nutrition, Bondy, France

REFERENCES:
- [Derived] Valensi P, Barber-Chamoux N, Rezki A, Lambert C, Pereira B, Duale C, Delmas D, Duclos M. Effects of single and multiple sessions of lower body diastole-synchronized compressions using a pulsating pneumatic suit on endothelium function and metabolic parameters in patients with type 2 diabetes: two controlled cross-over studies. Cardiovasc Diabetol. 2022 Dec 22;21(1):286. doi: 10.1186/s12933-022-01710-6. PMID 36550568